CLINICAL TRIAL: NCT03766555
Title: Microwave Ablation Versus Liver Resection For Early Hepatocellular Carcinoma in Patients With Borderline Liver Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Charing Chong, MD, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016.205
Record Dates: First submitted 2018-07-16; First posted 2018-12-06 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma; Hepatectomy; Microwave Ablation; Local Ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hepatectomy

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized study to be conducted in an academic hospital with a specialized hepato-biliary team. The principal investigator and other members within the team will perform patient selection and recruitment of this study according to the inclusion and exclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microwave Ablation (Experimental): Microwave ablation (MWA) will be performed in patients randomized to this arm.
  Interventions: Procedure: Microwave ablation
- Liver Resection (Active Comparator): Liver resection will be performed in patients randomized to this arm.
  Interventions: Procedure: Liver resection

INTERVENTIONS:
Procedure: Microwave ablation — Microwave ablation will be performed in operation theatre under general anesthesia via laparoscopic or open approach according to the tumors' locations. In case of open approach, it will be done via a right subcostal incision with possible upper midline extension was necessary. After diagnostic laparoscopy in laparoscopic approach and exploratory laparotomy in open approach to exclude the presence of extra-hepatic disease, operative ultrasound (Aloka, Tokyo, Japan) will be performed to exclude preoperatively undetected lesion; guide insertion of the microwave applicator; and monitor the whole ablation process. Surrounding organs were cooled by constant irrigation of ice-cold saline to prevent thermal injury. The ablation will be carried out according to the standard protocol with the aim to create a 1cm ablation margin around the tumor. The insertion track will be burnt after ablation in order to prevent bleeding and tumor seeding.
  Arms: Microwave Ablation
Procedure: Liver resection — Liver resection will be performed as described previously. Liver parenchymal transection would be performed with CUSA (cavitron ultrasonic surgical aspirator) and TissueLink (a radiofrequency saline-linked dissecting sealer) in both arms. Vascular staplers would be used to divide major vascular pedicles. Fibrin glue (Tisseel) spray would be applied to the parenchymal cut surface of the liver before closure of abdomen.
  Arms: Liver Resection

SUMMARY:
We propose a randomized controlled study to compare the treatment efficacy of microwave ablation to liver resection for hepatocellular carcinoma (HCC) in patients with borderline liver function.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a common cancer and is diagnosed at an earlier stage and with increasing frequency because of the wider implementation of screening programs. Whether liver resection or local ablation should be the first-line treatment in early HCC remains a hot topic for debate. Both are regarded as acceptable curative treatment for early HCC in many international guidelines. Underlying liver function is the key in treatment selection. The general consensus is that liver resection should be the treatment of choice in patients with good liver function while local ablation should be considered in patients with poor liver function. There exists a group of patients with apparently good liver function that harbor significant liver cirrhosis which is not easily picked up by the current assessment or scoring systems. Liver resection in this group of patients is burdened by potentially life-threatening complications and the overall survival is limited by their underlying liver cirrhosis. This is particularly important in early HCC as local ablation is another curative treatment option. In order to improve the prognosis of patients with early HCC, it is important to identify (1) patients with liver dysfunction to the extend that the risk of liver resection will outweigh the survival benefit it provides; (2) the best ablative method for HCC.

The investigators propose to carry out a prospective randomized controlled study to compare the treatment outcome of microwave ablation with liver resection in patients with borderline liver function whose HCC that are amendable to both liver resection and microwave ablation.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* HCC amendable for both MWA and liver resection
* Liver function of ALBI Grade 2
* Tumour size </= 5cm
* Absence of extrahepatic metastasis
* Absence of radiology evidence of major vascular or bile duct invasion

Exclusion Criteria:

* Informed consent not available
* Patients with ALBI 3, Child-Pugh B or above
* Multifocal tumour
* Presence of portal vein or hepatic artery thrombosis
* Anticipation of concomitant procedures
* Emergency hepatectomy
* Ruptured HCC
* Patients with chronic renal failure
* Pregnant female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2018-05-21 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  The primary outcome of this study is the overall survival

SECONDARY OUTCOMES:
Disease-free survival | 5 years
  Disease-free survival
Recurrence rate | 5 years
  Liver cancer recurrence rate
Morbidity rate | 1 year
  Morbidity rate
Hospital stay | 1 year
  Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Charing CN Chong, MBChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- See also: Hong Kong Hospital Authority. Hong Kong Cancer Registry. 2012. — http://www3.ha.org.hk/cancereg/pdf/overview/Summary%20of%20CanStat%202012.pdf